CLINICAL TRIAL: NCT02741063
Title: Oxytocin Effect on Attentional Bias Towards Emotional Expression Faces in Individuals With High and Low Autistic Traits: A Functional Magnetic Resonance Imaging (fMRI) Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Keith Kendrick, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UESTC-neuSCAN-19
Record Dates: First submitted 2016-03-30; First posted 2016-04-18 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: oxytocin; attentional bias; Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- high autistic and oxytocin group (Experimental): subject with high ASQ scores will receive oxytocin treatment
  Interventions: Behavioral: screen high autistic subjects; Drug: oxytocin
- low autistic and oxytocin group (Experimental): subject with low ASQ scores will receive oxytocin treatment
  Interventions: Behavioral: screen low autistic subjects; Drug: oxytocin
- high autistic and placebo group (Placebo Comparator): subject with high ASQ scores will receive placebo treatment
  Interventions: Behavioral: screen high autistic subjects; Drug: placebo
- low autistic and placebo group (Placebo Comparator): subject with low ASQ scores will receive placebo treatment
  Interventions: Behavioral: screen low autistic subjects; Drug: placebo

INTERVENTIONS:
Behavioral: screen low autistic subjects — screen subjects with low ASQ score
  Arms: low autistic and oxytocin group; low autistic and placebo group
Behavioral: screen high autistic subjects — screen subjects with high ASQ score
  Arms: high autistic and oxytocin group; high autistic and placebo group
Drug: oxytocin — intranasal administration of oxytocin (24 IU)
  Arms: high autistic and oxytocin group; low autistic and oxytocin group
Drug: placebo — intranasal administration of placebo (24 IU)
  Arms: high autistic and placebo group; low autistic and placebo group

SUMMARY:
to investigate whether oxytocin alter attentional bias towards emotional expression faces in individuals with high and low autistic traits, and the brain mechanism of this effect

DETAILED DESCRIPTION:
In the present study, investigator plan to use a double-blind, between-subject placebo controlled design.Firstly, all healthy male subjects' autistic trait levels will be assessed by the Autism Spectrum Quotient (ASQ) and only subjects with higher or lower ASQ score will be recruited in the next experiment and divided into high and low subgroup. Then, subjects are randomly assigned to receive either intranasal administration of oxytocin (24 IU) or placebo. 45 min later, subject need to complete an attentional bias task named rapid serial visual presentation (RSVP) task in fMRI scanner.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* history of head injury;
* claustrophobia;
* medical or psychiatric illness.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
attentional bias toward emotional expression faces | 1 hour
  attentional bias was measured by the accuracy of each emotional faces in the RSVP task

SECONDARY OUTCOMES:
brain activity during RSVP task | 1 hour
  brain activity was measured by the fMRI scanner

CONTACTS AND LOCATIONS:
Overall Officials: Keith Kendrick, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- China, Sichuan, Chengdu, Sichuan, China